CLINICAL TRIAL: NCT02157155
Title: The Role of ATGL and G0/G1 Switch Gene Complex in Lipopolysaccaride (LPS) Induced Ketosis - a Controlled, Randomised, Clinical Experimental Study
Brief Title: A Study of Intracellular Signaling in Muscle and Fat Cells During Ketosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-10-72-98-14
Record Dates: First submitted 2014-05-23; First posted 2014-06-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2014-06

CONDITIONS: Ketoacidosis; Diabetes Mellitus Type 1
MeSH Terms: conditions — Ketosis; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Insulin reduction and mimic infection with LPS
  Interventions: Biological: LPS
- Control (No Intervention): Normal insulin and no LPS

INTERVENTIONS:
Biological: LPS — LPS is endotoxin from gram negative bacteria. It is used scientifically to mimic infection lasting 4-8 hours.
  Arms: Intervention

SUMMARY:
Hypothesis

1. To define whether stimulation of ATGL and suppression of G0/G1 switch gene occur in the initial phases of diabetic ketoacidosis and thus can be identified as the primary mechanisms behind this life threatening condition.
2. Make a human model for studying ketoacidosis.

The investigators plan to reduce in their regular insulin over night. In the morning we administer endotoxin, which together with a relative lack of insulin will initiate ketogenesis - a state of ketoacidosis. On another occasion strict glycemic control is imposed by means of intravenous insulin. The testing is done two separate days with at least 3 weeks in between and patients are admitted to hospital the evening before the day of testing. The investigators use isotopic tracers to determine metabolic fluxes and analyse fat (ATGL, G0/G1 switch gene) and muscle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1
* 19 < BMI < 26
* minimal or negative C-peptide
* written consent

Exclusion Criteria:

* Severe comorbidity
* regular medication apart from insulin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Insulin signaling expressed as a CHANGE in phosphorylation of intracellular target proteins and CHANGE in mRNA expression of target genes in muscle- and fat-tissue. | Muscle and fat biopsies obtained on each study day (arm): t1= 6.45 (-75min) am t2=11.15 (195min) am t3= 12.30 pm (270min)
  Change in phosphorylation of target proteins and messenger RNA (mRNA) expression of target genes assessed with western blotting technique.

SECONDARY OUTCOMES:
Change in Intracellular markers of lipid metabolism in muscle- and fat tissue biopsies | Muscle and fat biopsies obtained on each study day (arm): t1= 6.45 am (-75min) t2=11.15 (195min) am t3= 12.30 pm (270min)
  Muscle and fat at t1 and t2. Muscle biopsy at t3. Intracellular markers are assessed by western blotting.
Metabolism | Change in glucose, fat and protein metabolism between study days and during each study day
  Change in glucose, fat and protein metabolism assessed by tracer kinetics on every study day (specific times below) and by indirect calorimetry. [3H 3]Glucose tracer from t=0 - 360min. Palmitic acid tracer from t=165min - 360min. Urea tracer from 0min - 240min. amino acid tracer from 60 min - 360 min.
Cytokines and stress hormones | In basal period t=0-240 minutes and in clamp period t=240-390 minutes
  Measurement of immune response to endotoxin and hypoinsulinaemia. Estimating the whole body stress during ketoacidosis and pre ketoacidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mads Svart, MD, Principal Investigator — Aarhus University / Aarhus University Hospital; Niels Møller, MD, Study Chair — Aarhus University / Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Andreasen AS, Krabbe KS, Krogh-Madsen R, Taudorf S, Pedersen BK, Moller K. Human endotoxemia as a model of systemic inflammation. Curr Med Chem. 2008;15(17):1697-705. doi: 10.2174/092986708784872393. PMID 18673219
- [Background] Zimmermann R, Strauss JG, Haemmerle G, Schoiswohl G, Birner-Gruenberger R, Riederer M, Lass A, Neuberger G, Eisenhaber F, Hermetter A, Zechner R. Fat mobilization in adipose tissue is promoted by adipose triglyceride lipase. Science. 2004 Nov 19;306(5700):1383-6. doi: 10.1126/science.1100747. PMID 15550674
- [Background] Bezaire V, Mairal A, Ribet C, Lefort C, Girousse A, Jocken J, Laurencikiene J, Anesia R, Rodriguez AM, Ryden M, Stenson BM, Dani C, Ailhaud G, Arner P, Langin D. Contribution of adipose triglyceride lipase and hormone-sensitive lipase to lipolysis in hMADS adipocytes. J Biol Chem. 2009 Jul 3;284(27):18282-91. doi: 10.1074/jbc.M109.008631. Epub 2009 May 11. PMID 19433586
- [Background] Haemmerle G, Lass A, Zimmermann R, Gorkiewicz G, Meyer C, Rozman J, Heldmaier G, Maier R, Theussl C, Eder S, Kratky D, Wagner EF, Klingenspor M, Hoefler G, Zechner R. Defective lipolysis and altered energy metabolism in mice lacking adipose triglyceride lipase. Science. 2006 May 5;312(5774):734-7. doi: 10.1126/science.1123965. PMID 16675698
- [Background] Schweiger M, Schreiber R, Haemmerle G, Lass A, Fledelius C, Jacobsen P, Tornqvist H, Zechner R, Zimmermann R. Adipose triglyceride lipase and hormone-sensitive lipase are the major enzymes in adipose tissue triacylglycerol catabolism. J Biol Chem. 2006 Dec 29;281(52):40236-41. doi: 10.1074/jbc.M608048200. Epub 2006 Oct 30. PMID 17074755
- [Background] Yang X, Lu X, Lombes M, Rha GB, Chi YI, Guerin TM, Smart EJ, Liu J. The G(0)/G(1) switch gene 2 regulates adipose lipolysis through association with adipose triglyceride lipase. Cell Metab. 2010 Mar 3;11(3):194-205. doi: 10.1016/j.cmet.2010.02.003. PMID 20197052
- [Background] Nielsen TS, Vendelbo MH, Jessen N, Pedersen SB, Jorgensen JO, Lund S, Moller N. Fasting, but not exercise, increases adipose triglyceride lipase (ATGL) protein and reduces G(0)/G(1) switch gene 2 (G0S2) protein and mRNA content in human adipose tissue. J Clin Endocrinol Metab. 2011 Aug;96(8):E1293-7. doi: 10.1210/jc.2011-0149. Epub 2011 May 25. PMID 21613358
- [Background] Burge MR, Garcia N, Qualls CR, Schade DS. Differential effects of fasting and dehydration in the pathogenesis of diabetic ketoacidosis. Metabolism. 2001 Feb;50(2):171-7. doi: 10.1053/meta.2001.20194. PMID 11229425
- [Background] Burge MR, Hardy KJ, Schade DS. Short-term fasting is a mechanism for the development of euglycemic ketoacidosis during periods of insulin deficiency. J Clin Endocrinol Metab. 1993 May;76(5):1192-8. doi: 10.1210/jcem.76.5.8496310.
- [Background] West MA, Heagy W. Endotoxin tolerance: A review. Crit Care Med. 2002 Jan;30(1 Supp):S64-S73. PMID 11891406
- [Background] Sanchez-Cantu L, Rode HN, Christou NV. Endotoxin tolerance is associated with reduced secretion of tumor necrosis factor. Arch Surg. 1989 Dec;124(12):1432-5; discussion 1435-6. doi: 10.1001/archsurg.1989.01410120082016. PMID 2589967
- [Background] Cahill GF Jr. Fuel metabolism in starvation. Annu Rev Nutr. 2006;26:1-22. doi: 10.1146/annurev.nutr.26.061505.111258. PMID 16848698
- [Derived] Lauritzen ES, Svart MV, Voss T, Moller N, Bjerre M. Impact of Acutely Increased Endogenous- and Exogenous Ketone Bodies on FGF21 Levels in Humans. Endocr Res. 2021 Feb;46(1):20-27. doi: 10.1080/07435800.2020.1831015. Epub 2020 Oct 19. PMID 33074729
- [Derived] Svart MV, Rittig N, Kampmann U, Voss TS, Moller N, Jessen N. Metabolic effects of insulin in a human model of ketoacidosis combining exposure to lipopolysaccharide and insulin deficiency: a randomised, controlled, crossover study in individuals with type 1 diabetes. Diabetologia. 2017 Jul;60(7):1197-1206. doi: 10.1007/s00125-017-4271-x. Epub 2017 Apr 7. PMID 28389705